CLINICAL TRIAL: NCT02908503
Title: Vaginal Film Administration and Placement Study: FLAG
Acronym: FLAG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Principal Investigator, Sharon Hillier, Professor, University of Pittsburgh
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: PRO16010551
Record Dates: First submitted 2016-08-15; First posted 2016-09-21 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2018-07

CONDITIONS: Healthy Women

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 x 2 inch PVA based film (Other): 1 x 2 inch polyvinyl acetate (PVA) based vaginal film
  Interventions: Other: Placebo Film
- 2 x 2 inch PVA based film (Other): 2 x 2 inch polyvinyl acetate (PVA) based vaginal film
  Interventions: Other: Placebo Film
- 1 x 2 cellulose based film (Other): 1 x 2 cellulose based vaginal film
  Interventions: Other: Placebo Film
- 2 x 2 cellulose based film (Other): 2 x 2 cellulose based vaginal film
  Interventions: Other: Placebo Film

INTERVENTIONS:
Other: Placebo Film — placebo vaginal films

SUMMARY:
The purpose of this study is to evaluate use of four different vaginal films - two sizes and two textures. The vaginal films have no active ingredients or medications. Information will be gathered about each film (i.e. ease of insertion, proper placement, opinions about each). The results of this study will help investigators determine which type of vaginal film to use (and how to write product instructions) for future studies.

DETAILED DESCRIPTION:
All women will use all 4 products in a randomized study design with a crossover evaluation during 10 visits over two months. Visits will be scheduled when the participant is not menstruating/bleeding. The sequence of film use will be randomized. Study procedures will involve a screening visit (VISIT 1) during which a baseline cervicovaginal lavage will be collected and infections will be excluded. After randomization (VISIT 2) women will be given instructions and instructed to insert the first film. An external genital examination will be performed after the participant inserts the film to verify film placement. In the event a participant has difficulty placing the film, the study clinician may place the film for them. Following each film insertion, a questionnaire will be administered to obtain feedback regarding ease of administration. Thirty minutes after product insertion a clinician will visualize film placement in the vagina by speculum examination. Women will be counseled to avoid sexual activity or vaginal product usage before VISIT 3 scheduled for the following day. At visit 3 women will have a speculum examination to assess whether the film has completed disintegrated and a CVL sample will be collected. Women will be given an appointment for the next film insertion in 7-20 days. The general sequence of events will be repeated for each subsequent film. At the next visit (VISIT 4) women will insert the second film and have the same evaluation as visit 2. A CVL sample will be collected 24 hours later (VISIT 5). Women will be asked to return to insert another film 7-20 days later (VISIT 6) and a CVL sample will be collected the next day (VISIT 7). Women will receive the final film 7-20 days later (VISIT 8) and have the final CVL collection following film insertion the next day (VISIT 9). A final visit (VISIT 10) will be scheduled >14 days after visit 9. During this visit a CVL will be collected for glycomic and innate antiviral activity studies and an in depth interview will be conducted in order to gain insights into the role of film polymer and size on perceived ease of insertion across the four film types.

ELIGIBILITY:
Inclusion Criteria:

1. Female, Age 18-40
2. Able and willing to provide written informed consent to be screened for and enrolled in the study.
3. Able and willing to provide adequate locator information at screening.
4. HIV-uninfected based on documented testing performed in the previous 6 months or by study staff at screening.
5. In general good health as determined by the site clinician
6. Agree to abstain from any intravaginal or rectal product or device or penetration (including vaginal, anal, or oral sex, masturbation, or sex toys) between each film insertion and the collection of the CVL approximately 24 hours later. Agree to be sexually abstinent for 48 hours prior to the study visits (from enrollment to visit 10). Sexual activity in the 48 hours prior to screening is acceptable.
7. Willingness to undergo all study-related assessments and procedures, including multiple speculum examinations, and follow all other study-related procedures
8. At screening and enrollment, agrees not to participate in other research studies involving drugs, medical devices, or vaginal products while enrolled in this trial and to abstain from vaginal product usage with the exception of tampons over the study period.

Exclusion Criteria:

Women who meet any of the following criteria by participant report will be excluded from the study. Of note, the study is limited to premenopausal women with an intact uterus because the mucosal immune environment differs substantially between pre- and post- menopausal women. Therefore, inclusion of post-menopausal women would introduce heterogeneity into the population.

1. Previous participation in a vaginal film study where participant was randomized to use film (i.e. FAME 02; FAME 04). Note: If participant was randomized to the gel arm, then she would be potentially eligible for participation in FLAG.
2. Menopausal at screening (as defined as amenorrhea for one year or more without an alternative etiology)
3. Hysterectomy
4. Participant report of any of the following at screening:

   1. Known adverse reaction to any of the study products (ever)
   2. Known adverse reaction to latex (ever)
   3. Non- therapeutic injection drug use in the 12 months prior to screening
   4. Surgical procedure involving the pelvis in the 90 days prior to screening (includes dilation and curettage or evacuation, and cryosurgery; does not include cervical biopsy for evaluation of an abnormal pap smear or IUD placement)
   5. Participation in a drug, spermicide and/or microbicide study in the 30 days prior to screening or anticipated participation in an investigational drug study in the next 8 weeks
   6. Currently pregnant or pregnancy within 90 days prior to screening
   7. Lactating
   8. Use of a diaphragm, NuvaRing®, or spermicide for contraception 5.) Urogenital infection or suspected infection within 14 days of enrollment including: symptomatic candidiasis, trichomonas vaginalis, and symptomatic bacterial vaginosis; or cervical infection, including Neisseria gonorrhoeae (GC), Chlamydia trachomatis (CT), or mucopurulent cervicitis; syphilis; HSV lesions, or other sores (Note: participants seropositive for HSV without active lesions will not be excluded); acute pelvic inflammatory disease; urinary tract infection

6. Antibiotic or antifungal therapy (vaginal or systemic) within 7 days of enrollment

7. Menses or other vaginal bleeding at the time of enrollment* or expecting menses in the 5 days after enrollment.

*Note, for women with monthly cycles, every attempt will be made to enroll these participants in the first half of their menstrual cycle. Women who have vaginal bleeding at the scheduled Enrollment Visit may return at a different date to be re-examined and possibly enrolled provided they are still within the screening window (maximum of 30 days between screening and enrollment) and meet all criteria.

8. Any condition that, in the opinion of the Investigator, would preclude provision of consent, make participation in the study unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2016-07; Primary Completion 2017-02-14 (Actual); Study Completion 2017-02-14 (Actual)

PRIMARY OUTCOMES:
correct insertion of vaginal films | approximately 2 months
  assessed by examination
ease of insertion of vaginal film | approximately 2 months
  assessed by questionnaire

SECONDARY OUTCOMES:
experience prior to film insertion | approximately 2 months
  as assessed by participant interviews
glycome/innate anti-HIV activity evaluation | approximately 2 months
  laboratory testing including cervicovaginal lavage
experience during film insertion | approximately 2 months
  as assessed by participant interviews
experience after film insertion | approximately 2 months
  as assessed by participant interviews

CONTACTS AND LOCATIONS:
Overall Officials: Sharon L Hillier, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- Magee-Womens Hospital of UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No